CLINICAL TRIAL: NCT06116734
Title: Open-label, Randomized Comparative Study to Assess Biosimilar Pegfilgrastim Versus Biosimilar Filgrastim in Patients With Multiple Myeloma and Lymphoma Post Autologous Hematopoietic Stem Cell Transplantation
Brief Title: Lapelga vs Gastrofil
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: Apobiologix. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1233770
Record Dates: First submitted 2023-09-19; First posted 2023-11-03 (Actual); Last update posted 2023-11-03 (Actual); Status verified 2023-10

CONDITIONS: Multiple Myeloma; Lymphoma; Engagement, Patient; Febrile Neutropenia
MeSH Terms: conditions — Multiple Myeloma; Lymphoma; Patient Participation; Febrile Neutropenia | interventions — TKN732

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Biosimilar pegfilgrastim (Experimental): Day +5 of cell infusion: Biosimilar pegfilgrastim or Lapelga™ (one dose)
  Interventions: Drug: Lapelga
- Biosimilar filgrastim (Active Comparator): Day +5 of cell infusion: Biosimilar filgrastim or Grastofil® (one dose for 5 days)
  Interventions: Drug: Grastofil®

INTERVENTIONS:
Drug: Grastofil® — On day 5 after the hemopoietic stem cell transplant, one subcutaneous injection for 5 days
  Other Names: biosimilar filgrastim
  Arms: Biosimilar filgrastim
Drug: Lapelga — On day 5 after the hemopoietic stem cell transplant, one subcutaneous injection
  Other Names: biosimilar pegfilgrastim
  Arms: Biosimilar pegfilgrastim

SUMMARY:
This study is examining one-time injection of biosimilar pegfilgrastim compared with multiple injection biosimilar filgrastim post autologous hematopoietic stem cell transplantation. Study aims to compare biosimilar pegfilgrastim - LaPelga and biosimilar filgrastim -Gastrofil to see if they are similar in efficacy in terms of neutrophil engraftment, limited adverse effects, and more convenience to our patients, with potential cost savings.

DETAILED DESCRIPTION:
This will be a prospective open randomized controlled study. The study will be conducted in the inpatient setting at the London Health Sciences Centre (LHSC) in London, ON, and Windsor Metropolitan Hospital (WMH) in Windsor, ON. The objective of the study is to assess if biosimilar Peg-filgrastim similar is non-inferior to biosimilar filgrastim (LaPelga versus gastrofil) in terms of neutrophil engraftment in autologous transplant patients with lymphoma and multiple myeloma.

Current clinical practice uses a risk-adapted approach where we use originator filgrastim - Neupogen starting on day 5 for patients who are aged 60 or greater, infusion of stem cells with a CD34 count less than or equal 3 x 10^6/kg, prior episodes of febrile neutropenia, or at the provider's clinical discretion. For the purposes of the trial, patients will be randomized to LaPelga versus gastrofil arm directly and will initiate assigned treatment at day+5 of autologous transplant.

Both LHSC and WMH have qualified investigators (hematologists or other qualified clinicians. The study will start only after receipt of regulatory and ethics approval. Screening investigations on patients will be done only after the signing of written informed consent.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be able and willing to give written informed consent prior to any study related procedures
* Patients with a diagnosis of multiple myeloma or lymphoma who are eligible for autologous stem cell transplant
* All adult patients aged 18 to 75 years
* All patients admitted to LHSC for autologous peripheral blood stem cell transplant receiving peripheral blood stem cell infusions at LHSC and post-transplant care at either LHSC or WMH.
* Of the patients who are admitted for autologous stem cell transplant, the patients that meet the risk adapted approach for GSCF will be included in the study. The risk adapted criteria are aged 60 or greater, infusion of stem cells with a CD34 count less than or equal 3 x 10^6/kg, prior episodes of febrile neutropenia, or at the providers clinical discretion
* Conditioning chemotherapy as per usual clinical practice

Exclusion Criteria:Patients satisfying the above inclusion criteria but with the following contraindications (prior to randomization) will be excluded from the study:

* Any clinical contraindications to filgrastim, e.g. hypersensitivity to G-CSF or E. coli-derived proteins
* Pain requiring opioids with use of filgrastim during mobilization of autologous stem cells.
* Unable or not willing to provide written consent

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2023-11-01 (Estimated); Primary Completion 2024-11-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
Engraftment | 11 days
  •Compare duration of neutropenia both in terms of absolute neutrophil count (ANC) <0.5 · 109 /l and of days to reach an ANC >0.5 · 109t between LaPelga versus gastrofil initiated at day 5 in patients with multiple myeloma or lymphoma post autologous transplant who meet the risk adapted criteria (age greater or equal to 60; prior episode of neutropenia and CD34 count of less than or equal to 3 X 10^6/kg cells infused)

SECONDARY OUTCOMES:
AE | 30 days
  * Clinically significant infections (CTCAE v 5, Infections, grade 2 or higher)
  * Grade and duration of mucositis (CTCAE v 5, mucositis oral and diarrhea, any grade)

CONTACTS AND LOCATIONS:
Overall Officials: Shona Philip, MD, Principal Investigator — London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's